CLINICAL TRIAL: NCT07069621
Title: Positive Parenting Program for Attention Deficit Hyperactivity Disorder: Maternal Perspective Shifts and Child Behavior Problems Reduction in a Clinical Trial
Brief Title: Triple P forADHD Children's Mothers, Education of Behavioral Problems, and Change in Mothers' Attitude
Acronym: (ADHD)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Palestine Polytechnic University (Other)
Responsible Party: Principal Investigator, Nadia Amro, D Nadia Amro,lecturer at Palestine Polytechnique university, Palestine Polytechnic University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: R-2024/A/131/N
Record Dates: First submitted 2025-06-21; First posted 2025-07-17 (Actual); Results first posted 2026-01-29 (Actual); Last update posted 2026-01-29 (Actual); Status verified 2026-01

CONDITIONS: ADHD, Predominantly Hyperactive - Impulsive; Behavior Problems, Child; ADHD - Attention Deficit Disorder With Hyperactivity; Healthy Adult Females; Competence; Positive Parenting
Keywords: sense of competency,mothers,ADHD,Behavioral problems; child; parenting attitudes; triple p
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity; Mental Disorders

STUDY DESIGN:
Intervention Model Description: One group received the Triple P program
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mothers of children with ADHD and with children with ADHD aged 6-12 years (Experimental): Had the Triple P sessions
  Interventions: Behavioral: Triple p level parenting program
- control (No Intervention): Did not receive triple p

INTERVENTIONS:
Behavioral: Triple p level parenting program — An evidence-based program with self-agency strategies enhances trust and confidence in managing children's ADHD behaviors
  Arms: Mothers of children with ADHD and with children with ADHD aged 6-12 years

SUMMARY:
The goal of this clinical trial is to investigate whether the Triple P program will reduce behavioral problems for ADHD children, improve mothers' sense of competency, and improve their attitudes

The main questions it aims to answer are:

1 . What is the feasibility and cultural acceptability of implementing the Triple P program within the Palestinian context? 2. Does the Triple P program promote positive attitudes towards managing ADHD among mothers in Palestine? 3. How does the Triple P program affect the maternal sense of competency among mothers in Palestine? 4. Does the Triple P program delivery affect reducing children's ADHD behavioural symptoms?

Participants :

took the triple p strategies, and the control will not Outcome measures will be evaluated pre- and post-intervention

DETAILED DESCRIPTION:
Mothers of children with ADHD are included; children with other mental health disorders or combined types of autism are excluded. The sample was taken from mental health clinics with children diagnosed with ADHD, aged 6-12 years old.

ELIGIBILITY:
The inclusion criteria:

1. having a child aged 6 - 13 years with an ADHD diagnosis
2. attending a child mental health clinic
3. No participation with another professional agency to receive parental support for mothers.

The exclusion criterion :

1. having a child with ADHD combined with neurological disorders
2. known medical conditions, severe aggression, intellectual disability, psychosis, and bipolar disorder.
3. children with ADHD older than 12 or younger than 6 years

Ages: 6 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 67 (Actual)
Dates: Start 2023-07-25 (Actual); Primary Completion 2024-08-30 (Actual); Study Completion 2024-08-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Nadia A Amro, phd, Principal Investigator — AAUP; Nadia A Amro, phd, Principal Investigator — Palestine Polytechnic University
Locations (1):
- Child Mental Health Clinic, Hebron, Palestinian Territories

IPD SHARING:
Plan to Share IPD: Yes
the whole process sesign prtocol ,data collection can be siscussed
Supporting Information: Study Protocol, ICF
Time Frame: one year
Access Criteria: any way of contact
URL: https://www.triplep.net/glo-en/home/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: subjects were recruited from a governmental child mental health clinic
Pre-assignment Details: files were searched for possible matched inclusion criteria
Groups:
- INTERVENTION: Mothers of children with ADHD and with children with ADHD aged 6-12 years:Had the Triple P sessions
- Control: Mothers of children with ADHD and with children with ADHD aged 6-12:Did not receive triple p
Period: Intervention
Arm/Group | INTERVENTION | Control
Started | 33 | 31
Completed | 33 | 31
Not Completed | 0 | 0
Period: 13 Months
Arm/Group | INTERVENTION | Control
Started | 33 | 31
Completed | 33 | 31
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Mothers of ADHD children
Groups:
- INTERVENTION: Group of intervention:Mothers of children with ADHD and with children with ADHD aged 6-12 years recieved Triple P
- CONTROL: Mothers of children with ADHD and with children with ADHD aged 6-12 years did not recieve triple p
- Total: Total of all reporting groups
Arm/Group | INTERVENTION | CONTROL | Total
Number analyzed (Participants) | 33 | 31 | 64
Age, Categorical [Count of Participants; unit: Participants] — mothers of children
  Participants
    <=18 years | 0 | 0 | 0
    Between 18 and 65 years | 33 | 31 | 64
    >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants] — mothers of ADHD children Population: non
  Participants
    Female | 33 | 31 | 64
    Male | 0 | 0 | 0
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Count of Participants; unit: Participants]
  Palestine | 33 | 31 | 64
The Parenting Sense of Competence Scale PSOC [Mean (Standard Deviation); unit: units on a scale] — The Parenting Sense of Competence (PSOC) scale (Gibaud-Wallston & Wandersman, 1978) is a 17-item self-report instrument assessing parents' perceived competence in their parenting role. Each item is rated on a 6-point Likert scale (1 = strongly disagree to 6 = strongly agree) . Possible Score Range: 16 to 96 High Total Score (e.g., 75+): Generally indicates a positive, adaptive parenting self-concept.
  Low Total Score (e.g., below 50): Indicates significant parenting distress and is a red flag for needed support.
  * with higher scores indicating greater parenting efficacy and satisfaction"
  units on a scale | 63.44 (9.67) | 65.03 (8.81) | 64.22 (9.44)
The Parenting Scale PS [Mean (Standard Deviation); unit: units on a scale] — The Parenting Scale a brief 7-item parent-report tool to assess dysfunctional parenting discipline. measures Laxness 4 items: Reflects permissive discipline and inconsistent enforcement of rules.
  Overreactivity 3 items: Captures harsh, irritable, or angry responses to child misbehavior.
  Each item is rated on a 7-point Likert-type scale, ranging from 1(effective discipline) to 7(ineffective discipline).
  Laxness score: Mean of 4 items (range: 1.0-7.0) higher scores mean worse it should not exceed 4 Over reactivity score: Mean of 3 items (range: 1.0-7.0) higher scores are worse,cutoff is 4
  units on a scale | 3.0 (0.87) | 3.8 (0.76) | 3.39 (0.81)
Strengths and Difficulties Questionnaire (SDQ) Subscales [Mean (Standard Deviation); unit: units on a scale] — The SDQ is a behavioral screening questionnaire assessing child emotional and behavioral difficulties. It contains subscales measuring Emotional Problems, Conduct Problems, Hyperactivity, Peer Problems, and Prosocial Behavior. Each subscale score ranges from 0 to 10, with higher scores indicating greater difficulties except for Prosocial Behavior, where higher scores indicate better social behavior. Scores are reported as means with standard deviations. Total difficulties score ranges from 0 to 40, with higher scores indicating more severe behavioral problems.
  units on a scale | 19.78 (5.56) | 21.32 (6.09) | 20.61 (5.82)

OUTCOME MEASURES:

1. Primary Outcome: SDQ: Strengths and Difficulties Questionnaire SDQ
Description: The Strengths and Difficulties Questionnaire (SDQ) is a validated behavioral screening tool that assesses emotional and behavioral difficulties in children through 25 items grouped into five subscales: Emotional Symptoms, Conduct Problems, Hyperactivity/Inattention, Peer Relationship Problems, and Prosocial Behavior. Each subscale includes 5 items scored from 0 to 2, resulting in subscale scores ranging from 0 to 10. Higher scores on the first four subscales indicate greater difficulties, while higher scores on the Prosocial Behavior subscale reflect better social functioning. A Total Difficulties Score (the lowest is 0 and the highest is 40) is calculated by summing the four difficulties subscales, with higher scores indicating more behavioral problems. Scores are reported as mean ± standard deviation, with higher total or subscale scores indicating worse outcomes for difficulties and better outcomes for prosocial behavior (Goodman, 1997; Stone et al., 2010)
Time Frame: Pre (Baseline) intervention and Post (12 months)
Population: mothers of ADHD children
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Intervention: had the triple p
- Control: did not triple p
Arm/Group | Intervention | Control
Number analyzed (Participants) | 33 | 31
score on a scale
  hyperactivity pre | 8.22 (1.98) | 7.71 (2.04)
  hyperactivity post | 6.78 (2.70) | 7.97 (2.01)
  Prosocial Pre | 7.47 (2.29) | 6.42 (2.81)
  prosocial Post | 7.72 (2.20) | 6.19 (2.57)
  SDQ-Peer Problems Pre | 4.38 (1.88) | 3.84 (1.51)
  SDQ-Peer Problems (Post) | 3.97 (1.71) | 3.90 (1.76)
  SDQ-Total Score Pre | 19.78 (5.56) | 21.32 (6.09)
  SDQ-Total Score Post | 19.28 (6.71) | 21.52 (5.54)

2. Secondary Outcome: Parenting Scale
Description: The Parenting Scale - Short Version is a brief 7-item parent-report tool designed to assess dysfunctional parenting discipline styles. It measures two core constructs:
  Laxness (4 items): Reflects permissive discipline and inconsistent enforcement of rules.
  Overreactivity (3 items): Captures harsh, irritable, or angry responses to child misbehavior.
  Each item is rated on a 7-point Likert-type scale, ranging from 1 (effective discipline) to 7 (ineffective discipline). Scores are computed as follows:
  Subscale Scores:
  Laxness score: Mean of 4 items (range: 1.0-7.0) higher scores mean worse it should not exceed 4
  Over reactivity score: Mean of 3 items (range: 1.0-7.0) higher scores are worse , cutoff is 4
  Total Score: Mean of all 7 items (range: 1.0-7.0)
Time Frame: "Pre (Baseline)"intervention and "Post (12 months)")
Population: Mothers of ADHD children
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention | Control
Number analyzed (Participants) | 33 | 31
score on a scale
  Parenting Scale - Laxness (Pre) | 3.0 (1.2) | 3.8 (1.0)
  Parenting Scale - Laxness (Post) | 3.3 (1.4) | 3.9 (.9)
  Parenting Scale - Over reactivity (Pre) | 4.0 (1.3) | 3.9 (1.0)
  Parenting Scale - Over reactivity (Post) | 3.6 (1.3) | 3.7 (0.9)
  Parenting Scale - Total (Pre) | 3.77 (0.87) | 3.96 (0.76)
  Parenting Scale - Total (Post) | 3.22 (0.86) | 3.53 (0.63)

3. Secondary Outcome: PSOC: Parenting Sense of Competence PSOC Scale
Description: The Parenting Sense of Competence (PSOC) scale (Gibaud-Wallston & Wandersman, 1978) is a 17-item self-report instrument assessing parents' perceived competence in their parenting role. Each item is rated on a 6-point Likert scale (1 = strongly disagree to 6 = strongly agree) . Possible Score Range: 16 to 96
  Interpretation of Range:
  High Total Score (e.g., 75+): Generally indicates a positive, adaptive parenting self-concept.
  Low Total Score (e.g., below 50): Indicates significant parenting distress and is a red flag for needed support.
  * with higher scores indicating greater parenting efficacy and satisfaction"
Time Frame: "Pre (Baseline)"intervention and "Post (12 months)")
Population: Mothers of ADHD children
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Intervention: Mothers of children with ADHD and with children with ADHD aged 6-12 years :Had the Triple P sessions
Arm/Group | Intervention | Control
Number analyzed (Participants) | 33 | 31
score on a scale
  pre | 63.44 (6.97) | 65.03 (8.38)
  post | 68.28 (9.67) | 62.80 (8.81)

ADVERSE EVENTS:
Time Frame: 13 months, adverse events monitored but not found
Groups:
- Control: Mothers of children with ADHD and with children with ADHD aged 6-12 years: Did not receive Triple P
Arm/Group | Intervention | Control
All-Cause Mortality (participants affected / at risk) | 0/33 | 0/31
Serious Adverse Events (participants affected / at risk) | 0/33 | 0/31
Other Adverse Events (participants affected / at risk) | 0/33 | 0/31

LIMITATIONS AND CAVEATS:
First, the study used a pre-post design with no long-term follow-up, limiting insight into sustained effects. Second, the sample size was modest, affecting generalizability. Third, intervention delivery by a single researcher may have introduced social desirability bias. Lastly, data collection occurred during the Gaza conflict and lockdowns. Early termination leading to small numbers of subjects analyzed; Technical problems with measurement leading to unreliable or uninterpretable data.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2025-02-24): https://cdn.clinicaltrials.gov/large-docs/21/NCT07069621/Prot_SAP_002.pdf
  • Informed Consent Form (2023-04-30): https://cdn.clinicaltrials.gov/large-docs/21/NCT07069621/ICF_003.pdf